CLINICAL TRIAL: NCT02532335
Title: Study of the Effects of Obeticholic Acid on Farnesoid X Receptor Expression in Jejunum and on Gut Microbiota in Morbidly Obese Patients and Healthy Volunteers
Brief Title: Obeticholic Acid in Morbidly Obese Patients and Healthy Volunteers
Acronym: OCAPUSH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Hanns-Ulrich Marschall, Professor of Clinical Hepatology, Sponsor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OCAPUSH
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Obesity
Keywords: FXR; bile acids; FGF19; C4; gut microbiota; Pharmacodynamics of FXR activation in the small bowel
MeSH Terms: conditions — Obesity | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Morbid Obesity OCA (Active Comparator): Obeticholic acid 25 mg/day in three weeks
  Interventions: Drug: Obeticholic acid
- Morbid Obesity Placebo (Placebo Comparator): Obeticholic acid 25 mg/day matching placebo in three weeks
  Interventions: Drug: Obeticholic acid; Drug: Obeticholic acid placebo
- Healthy Volunteers OCA (Active Comparator): Obeticholic acid Obeticholic acid 25 mg/day in three weeks
  Interventions: Drug: Obeticholic acid
- Healthy volunteers Placebo (Placebo Comparator): Obeticholic acid 25 mg/day matching placebo in three weeks
  Interventions: Drug: Obeticholic acid; Drug: Obeticholic acid placebo

INTERVENTIONS:
Drug: Obeticholic acid — active drug
  Other Names: INT-747
Drug: Obeticholic acid placebo — matching placebo
  Other Names: INT-747 placebo
  Arms: Healthy volunteers Placebo; Morbid Obesity Placebo

SUMMARY:
OCAPUSH (EudraCT 2014-002313-33) is a double-blind placebo-controlled parallel-arms study of the effects of obeticholic acid on farnesoid X receptor expression in jejunum and on gut microbiota in morbidly obese patients and healthy volunteers. Obeticholic acid (OCA, 6-ethyl-chenodeoxycholic acid, INT-747) is a semi-synthetic derivative of the major human bile acid chenodeoxycholic acid and will be administered orally at a dose of 25 mg/day during three weeks to 20 morbidly obese patients awaiting Roux-en-Y gastric bypass and to 20 healthy volunteers. On the days before the first and after the last dose faeces and blood are sampled for the analyses of bile acids and the gut microbiota. On the day after the last dose a push-enteroscopy is performed in conscious sedation for biopsy taking in the jejunum.These procedures are repeated 6 month after surgery in the morbid obese patients. Inclusion criteria are male or female gender, 20-65 years of age and morbid obesity (BMI >35 kg/m2) eligible for bariatric surgery. Exclusion criteria are liver diseases other that fatty liver disease, other significant morbidity, medications known to interact with OCA, pregnancy, uncertainty about safe and reliable contraception, and problems to understand or adhere to the protocol. The primary objectives of this pharmacodynamic trial are the study of the effect of OCA on the expression of FXR in the jejunum and small intestinal permeability, and on fecal bile acids and gut microbiota. The secondary objectives are the study of the effects of OCA on the genome-wide FXR DNA binding sites (cistromics) with the global gene expression profile (transcriptomics) in human jejunum.

DETAILED DESCRIPTION:
Obeticholic acid will be administered orally at a dose of 25 mg/day during three weeks to 20 morbidly obese patients awaiting Roux-en-Y gastric bypass and to 20 healthy volunteers. On the days before the first and after the last dose faeces and blood are sampled for the analyses of bile acids and the gut microbiota. On the day after the last dose a push-enteroscopy is performed in conscious sedation for biopsy taking in the jejunum. These procedures are repeated 6 month after surgery in the morbid obese patients. Inclusion criteria are male or female gender, 20-65 years of age and morbid obesity (BMI >35 kg/m2) eligible for bariatric surgery. Exclusion criteria are liver diseases other that fatty liver disease, other significant morbidity, medications known to interact with OCA, pregnancy, uncertainty about safe and reliable contraception, and problems to understand or adhere to the protocol. The primary objectives of this pharmacodynamic trial are the study of the effect of OCA on the expression of FXR in the jejenum and small intestinal permeability, and on fecal bile acids and gut microbiota. The secondary objectives are the study of the effects of OCA on the genome-wide FXR DNA binding sites (cistromics) with the global gene expression profile (transcriptomics) in human jejunum.

ELIGIBILITY:
Inclusion Criteria:

Morbid obesity awaiting gastric bypass surgery, ≥35 kg/m2

Male subjects, pre-, and post-menopausal female subjects

Women of childbearing potential can only be included if a safe and reliable contraception is used, e.g., oral contraceptives

Patients eligible to laparoscopic bariatric surgery

Patients must give their signed and dated written consent to participate in this study based on written information of all pertinent aspects of the trial provided at least 24 hours before undertaking any trial related activity.

Exclusion Criteria:

Chronic liver disease other than NAFLD (viral hepatitis, autoimmune liver disease, hemochromatosis, homozygous alpha1-antitrypsin deficiency and Wilson disease)

Previous gastric or small bowel surgery

Inflammatory bowel disease

Uncontrolled diabetes mellitus (fasting blood glucose >6.7 mmol/L), hypothyroidism or hyperthyroidism, or other significant endocrine disease.

Pregnancy. A urine pregnancy test will be performed the day before start of medication. Women of childbearing potential can only be included if a safe and reliable contraception is used, e.g., oral contraceptives.

Elevations of transaminases (ALAT/ASAT) or alkaline phosphatase or bilirubin above 2xULN (upper limit of normal) the day before start of medication.

Other serious disease, including depressive disorders treated by medication

Patients who will not comply with the protocol.

Hypothyroidism, unless the subject is clinically euthyroid, receiving a stable dose thyroid hormone replacement therapy and serum TSH is within the normal range.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
ChIP-assay in biopsies as a measure of Activation of FXR-dependent genes in small intestine | Three weeks
  ChIP-assay in biopsies

SECONDARY OUTCOMES:
Shot-gun metagenomics as a measure of Impact of FXR activation on gut microbiota | Three weeks
  Shot-gun metagenomics

CONTACTS AND LOCATIONS:
Overall Officials: Hanns-Ulrich Marschall, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Hanns-Ulrich Marschall, Gothenburg
  - Sahlgrenska Academy, Gothenburg

IPD SHARING:
Plan to Share IPD: No